CLINICAL TRIAL: NCT04815213
Title: The Use of Expanded Mesenchymal Stromal Cells (MSC) in Premature Ovarian Failure (POF) in Adult Humans: Phase I Clinical Trial
Brief Title: The Use of Expandeded Mesenchymal Stromal Cells (MSC) in Premature Ovarian Failure (POF) in Adult Humans
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Hanan Jafar, Vice director/ Cell therapy center, University of Jordan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: POF.UJCTC
Record Dates: First submitted 2021-03-02; First posted 2021-03-24 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Premature Ovarian Failure
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MSCs Intravaginally (Experimental): Expanded autologous bone marrow-derived mesenchymal cells (BMMSCs), dose 20 million cells/ovary Inravaginally
  Interventions: Biological: expanded autologous bone marrow derived MSC Intravaginally
- MSCs Laparoscopic (Experimental): Expanded autologous bone marrow-derived mesenchymal cells (BMMSCs), dose 20 million cells/ovary Laparoscopic
  Interventions: Biological: expanded autologous bone marrow derived MSC Laporoscopic
- EV (Experimental): Extravascular vesicles (EV) injection
  Interventions: Biological: EV

INTERVENTIONS:
Biological: expanded autologous bone marrow derived MSC Intravaginally — Autologous bone marrow-derived mesenchymal cells (BMMSCs), dose 20 million cells/ovary
  Other Names: BM-MSc
  Arms: MSCs Intravaginally
Biological: expanded autologous bone marrow derived MSC Laporoscopic — Autologous bone marrow-derived mesenchymal cells (BMMSCs), dose 20 million cells/ovary
  Arms: MSCs Laparoscopic
Biological: EV — Extracellular vesicles injection
  Arms: EV

SUMMARY:
Autologous bone marrow-derived mesenchymal cells will be injected into patients diagnosed with premature ovarian failure

DETAILED DESCRIPTION:
MSCs in passage-2 culture will be washed with PBS and detached with trypsin/EDTA (0.25%). After that, the cells will be suspended at a density of 20×106 cells/ 2 ml normal saline and loaded into 3 ml sterile syringes.

The cells should be infused within 2 hours of release. Tests and follow up are to be monthly.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent
2. Married female, 18-38 years old
3. Diagnosis of premature ovarian insufficiency: At least two menopausal FSH levels (≥ 20 IU/L) and/or Primary or secondary amenorrhea at least for 6 months
4. Evidence of low ovarian reserve defined as: AMH < _0.3 ng/ML & FSH >20 IU/L, AFC < 4, and/or failure of prior attempts of assisted reproductive techniques due to limited ovarian response (poor responder).
5. Normal karyotype 46, XX.
6. Presence of at least one ovary
7. Normal thyroid function as evidence by normal serum Thyroid Stimulating Hormone (TSH) levels.
8. Agree to report any pregnancy to the research staff immediately.
9. Cooperative patient
10. Negative for infectious panel (HIV, HBV, HCV, and VDRL)

Exclusion Criteria:

1. Currently breast-feeding
2. Has a history of, or evidence of current malignancy
3. Major mental health disorder that precludes participation in the study
4. Current or recent (within the past 2 weeks) use of the following medications: Oral or systemic corticosteroids, Hormones (estrogen, progestins, oral contraceptives), Danazol, anticoagulants, herbal or botanical supplements with possible hormonal effects. Washout will be allowed.
5. Type I or Type II diabetes mellitus, or if receiving antidiabetic medications
6. Significant anemia (Hemoglobin <8 g/dL).
7. Untreated deep venous thrombosis, and/or pulmonary embolus
8. Known heart disease (New York Heart Association Class II or higher).
9. Known Liver disease (defined as Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT)>2 times normal, or total bilirubin >2.5 mg/dL).
10. Known Renal disease (defined as Blood urea nitrogen (BUN)>30 mg/dL or serum creatinine > 1.6 mg/dL).
11. Clinically active autoimmune condition

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Married female
Enrollment: 10 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 12 months
  Treatment adverse events are defined by any adverse event leading to hospitalization, organ failure or death

SECONDARY OUTCOMES:
Number of patients with enhanced hormonal profile, ovarian changes and endometrial changes | 12 months
  Efficacy will be measured comparing hormonal changes (FSH, LH, AMH, estradiol) in patients' blood on monthly intervals
Number of patients with positive ovarian changes | 12 months
  Patients ultrasounds of the ovaries will compare size and follicle numbers
Number of patients with increased endometrial thickness | 12 months
  Ultrasounds of uterus will be compared for endometrial thickness

CONTACTS AND LOCATIONS:
Overall Officials: Dr Abdalla Awidi, MD, Study Chair — Cell therapy center
Locations (1):
- Cell Therapy Center, University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No